CLINICAL TRIAL: NCT03226366
Title: Effect of Emergency Department Care Reorganization on Door-to-antibiotic Times for Sepsis (LDS SWARM)
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Ithan Peltan, Attending Physician, Intermountain Medical Center, Intermountain Health Care, Inc.
Other Study IDs: LDS SWARM
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Septic Shock; Sepsis
Keywords: door-to-antibiotic time; emergency department care; antimicrobial; care reorganization; severe sepsis; swarming
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — RsbA protein, Proteus mirabilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-implementation (intervention site): Adult patients age ≥18 years who received usual care after presenting to the ED of the intervention hospital with sepsis or septic shock between May 16, 2015 and April 15, 2016
- Post-implementation (intervention site): Adult patients age ≥18 years eligible to receive immediate evaluation by multidisciplinary team ("swarming") after presenting to the ED of the intervention hospital with sepsis or septic shock between May 16, 2016 and February 15, 2017
  Interventions: Other: Immediate evaluation by multidisciplinary team
- Pre-implementation (control site): Adult patients age ≥18 years who received usual care after presenting to the ED of a non-intervention study hospital with sepsis or septic shock between May 16, 2015 and April 15, 2016
- Post-implementation (control site): Adult patients age ≥18 years who received usual care after presenting to the ED of a non-intervention study hospital with sepsis or septic shock between May 16, 2016 and February 15, 2017

INTERVENTIONS:
Other: Immediate evaluation by multidisciplinary team — Simultaneous initial evaluation by the ED physician, nurse, and patient care associate
  Other Names: Swarming
  Groups: Post-implementation (intervention site)

SUMMARY:
Sepsis is a common syndrome resulting from a dysregulated response to infection. The timing of antibiotic initiation is an important determinant of outcomes for patients presenting to the emergency department with sepsis. The potential effect of care reorganization on very early care for sepsis is unknown. This study will investigate whether multidisciplinary coordination of the initial patient evaluation in the emergency department influences door-to-antibiotic time for septic patients.

DETAILED DESCRIPTION:
This is a retrospective cohort study of emergency department sepsis care before versus after implementation of a "swarming" model for simultaneous patient evaluation by multidisciplinary care providers. The analysis will use data from similar hospitals that did not change sepsis care organization during the study period to control for changes in sepsis care not resulting from the "swarming" intervention.

ELIGIBILITY:
Primary inclusion criteria:

* Adult patients age ≥18 years
* Presented to the ED of study hospital from May 16, 2015 to April 15, 2016 (pre-implementation cohort) or May 16 to November 15, 2016 (post-implementation cohort)
* Sepsis present in ED (Sequential Organ Failure Assessment [SOFA] score ≥2 points above baseline while in ED plus antibiotic initiation while in the ED)
* Triage acuity score 2-5

Inclusion criteria for supplemental sensitivity analyses:

* Presented to the ED of study hospital between May 16, 2015 and April 15, 2016 (pre-implementation cohort) or May 16, 2016 and February 15, 2017 (post-implementation cohort).
* Sepsis on presentation to ED, defined as initial Sequential Organ Failure Assessment (SOFA) score ≥2 points above baseline plus antibiotics initiation within 24 hours of ED arrival.

Overall exclusion criteria:

* Age <18 years
* No antibiotics within 24 hours of ED arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the ED with sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 3230 (Actual)
Dates: Start 2015-05-16 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2020-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ithan Peltan, MD, MSc, Principal Investigator — Intermountain Health Care, Inc.
Locations (4):
- United States (4):
  - Intermountain Medical Center, Murray, Utah
  - Riverton Hospital, Riverton, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Alta View Hospital, Sandy City, Utah

IPD SHARING:
Plan to Share IPD: Yes
In order to protect patient privacy and comply with relevant regulations, identified data will be unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.
Supporting Information: Study Protocol, CSR, Analytic Code

REFERENCES:
- [Result] Peltan ID, Bledsoe JR, Brems D, McLean S, Murnin E, Brown SM. Institution of an emergency department "swarming" care model and sepsis door-to-antibiotic time: A quasi-experimental retrospective analysis. PLoS One. 2020 May 5;15(5):e0232794. doi: 10.1371/journal.pone.0232794. eCollection 2020. PMID 32369531

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-implementation (Intervention Site): Adult patients age ≥18 years eligible to receive immediate evaluation by multidisciplinary team ("swarming") after presenting to the ED of the intervention hospital with sepsis or septic shock between May 16, 2016 and November 15, 2016
  Immediate evaluation by multidisciplinary team: Simultaneous initial evaluation by the ED physician, nurse, and patient care associate
- Post-implementation (Control Site): Adult patients age ≥18 years who received usual care after presenting to the ED of a non-intervention study hospital with sepsis or septic shock between May 16, 2016 and November 15, 2016
Period: Overall Study
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site)
Started | 911 | 495 | 1183 | 641
Completed | 911 | 495 | 1183 | 641
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site) | Total
Number analyzed (Participants) | 911 | 495 | 1183 | 641 | 3230
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (19.7) | 55.6 (19.6) | 59.9 (19.7) | 58.7 (20.4) | 57.6 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 474 | 251 | 687 | 377 | 1789
  Male | 437 | 244 | 496 | 264 | 1441
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 74 | 69 | 45 | 305
  Not Hispanic or Latino | 794 | 421 | 1114 | 596 | 2925
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 9 | 5 | 2 | 31
  Asian | 14 | 8 | 18 | 5 | 45
  Native Hawaiian or Other Pacific Islander | 30 | 12 | 12 | 13 | 67
  Black or African American | 25 | 15 | 6 | 4 | 50
  White | 827 | 451 | 1142 | 617 | 3037
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From ED Arrival to Administration of First Dose of Antibiotics
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site)
Number analyzed (Participants) | 911 | 495 | 1183 | 641
minutes | 173 (98) | 165 (95) | 169 (90) | 163 (85)
Statistical Analysis 1: Comparison: Pre-implementation (Intervention Site) vs Post-implementation (Intervention Site) vs Pre-implementation (Control Site) vs Post-implementation (Control Site); Differences-in-differences analysis using multivariable regression to estimate the change in emergency department (ED) door-to-antibiotic time after versus before intervention implementation at the intervention site adjusted for the change observed over the same time period at the control sites and for subject's age, sex, Elixhauser Comorbidity Score, initial systolic blood pressure, initial Glasgow Coma Scale score <14. initial temperature, ED triage acuity score, and ED arrival via ambulance; Test type: Superiority; p = 0.29, Regression, Linear; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-20.4 to 6.1] — Change in emergency department door-to-antibiotic time (minutes) based on adjusted differences-in-differences analysis

2. Secondary Outcome: Hospital Mortality
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site)
Number analyzed (Participants) | 911 | 495 | 1183 | 641
Participants | 19 | 7 | 23 | 11
Statistical Analysis 1: Comparison: Pre-implementation (Intervention Site) vs Post-implementation (Intervention Site) vs Pre-implementation (Control Site) vs Post-implementation (Control Site); Differences-in-differences analysis using multivariable regression to estimate the change in odds of hospital mortality after versus before implementation at the intervention site with adjustment for observed change in outcome over the same time period at the control sites as well as for subject's age, sex, Elixhauser Comorbidity Score, initial systolic blood pressure, an initial Glasgow Coma Scale score <14. initial temperature, ED triage acuity score, and arrival to the ED via ambulance; Test type: Superiority; p = 0.72, Regression, Logistic; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.25 to 2.61] — Odds ratio for hospital mortality after versus before intervention implementation based on adjusted differences-in-differences analysis

3. Secondary Outcome: ED Length of Stay
Description: Time (minutes) from ED arrival to ED departure
Time Frame: Up to 1 week
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site)
Number analyzed (Participants) | 911 | 495 | 1183 | 641
minutes | 280 (1143) | 265 (110) | 269 (108) | 261 (98)
Statistical Analysis 1: Comparison: Pre-implementation (Intervention Site) vs Post-implementation (Intervention Site) vs Pre-implementation (Control Site) vs Post-implementation (Control Site); Differences-in-differences analysis using multivariable regression to estimate the change in emergency department length of stay after versus before implementation at the intervention site with adjustment for the change observed over the same time period at the control sites as well as for subject's age, sex, Elixhauser Comorbidity Score, initial systolic blood pressure, an initial Glasgow Coma Scale score <14. initial temperature, ED triage acuity score, and arrival to the ED via ambulance; Test type: Superiority; p = 0.26, Regression, Linear; Mean Difference (Final Values) = -9.5, 95% CI 2-sided [-25.9 to 7.0] — Change in emergency department length of stay (minutes) after versus before intervention implementation based on adjusted differences-in-differences analysis

4. Secondary Outcome: Door-to-physician Evaluation Time
Description: Time (minutes) from subject's arrival in the ED until initial evaluation by a physician.
Time Frame: Up to 24 hours
Population: Time of physician initial patient evaluation was missing for a small number of participants in each group
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site)
Number analyzed (Participants) | 901 | 489 | 1164 | 624
minutes | 25 (18) | 23 (15) | 22 (24) | 20 (16)
Statistical Analysis 1: Comparison: Pre-implementation (Intervention Site) vs Post-implementation (Intervention Site) vs Pre-implementation (Control Site) vs Post-implementation (Control Site); Differences-in-differences analysis using multivariable regression to estimate the change in emergency department (ED) door-to-physician evaluation time after versus before implementation at the intervention site adjusted for the change observed over the same time period at the control sites and for subject's age, sex, Elixhauser Comorbidity Score, initial systolic blood pressure, initial Glasgow Coma Scale score <14. initial temperature, ED triage acuity score, and ED arrival via ambulance; Test type: Superiority; p = 0.55, Regression, Linear; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.3 to 1.8] — Estimated change in emergency department door-to-physician evaluation time (minutes) after versus before intervention implementation based on adjusted differences-in-differences analysis

ADVERSE EVENTS:
Time Frame: 1 year
Description: Intervention effects on hospital mortality and emergency department length of stay were evaluated as study outcomes. Other adverse events were not systematically collected given this was a retrospective study employing review of the electronic clinical record to evaluate a previously-implemented quality improvement initiative reordering of routine emergency department care for patients with sepsis.
Arm/Group | Pre-implementation (Intervention Site) | Post-implementation (Intervention Site) | Pre-implementation (Control Site) | Post-implementation (Control Site)
All-Cause Mortality (participants affected / at risk) | 19/911 | 7/495 | 23/1183 | 11/641
Serious Adverse Events (participants affected / at risk) | 0/911 | 0/495 | 0/1183 | 0/641
Other Adverse Events (participants affected / at risk) | 0/911 | 0/495 | 0/1183 | 0/641

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03226366/Prot_SAP_000.pdf